CLINICAL TRIAL: NCT03692325
Title: Safety and Efficacy of Nivolumab in Treating Oral Proliferative Verrucous Leukoplakia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-387
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Leukoplakia, Oral
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): * Nivolumab will be administered by IV infusion on Day 1 of each 28-day cycle
  * Treatment with the study drug will continue for a maximum of 4 cycles or until unacceptable toxicity or withdrawal of consent
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells.
  Other Names: Opdivo

SUMMARY:
This research study is studying an immunotherapy drug, as a possible treatment for oral proliferative verrucous leukoplakia (OPVL).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or combination of drugs to learn whether it works in treating a specific disease. "Investigational" means that the drug/s is being studied.

The purpose of this study is to evaluate effectiveness (how well the drug works) of nivolumab in treating OPVL and or prolonging the onset of possible malignancy.

Nivolumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells. Nivolumab has been demonstrated to activate the immune system to attack cancer cells in participants with different types of cancers. OPVL has a high risk for turning into cancer and the investigators are testing if nivolumab may help to shrink the white lesions in the participant's mouth and reduce cancer risk.

In November 2016, the Food and Drug Administration (FDA) approved nivolumab for the treatment of participants with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN). Squamous cell carcinoma is the kind of cancer that OPVL can transform into.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically confirmed oral proliferative verrucous leukoplakia (OPVL), as defined by: multifocal lesions (≥ 2) or contiguous lesions ≥ 3 cm or a single lesion ≥ 4 cm in largest diameter (at least one lesion with any degree of dysplasia). (Note: no restriction on the length of time that patients have had one or more existing lesions)
* Willing to provide blood and tissue from diagnostic biopsies
* Any smoking history is permitted. A history of prior or current tobacco use is not an exclusion criteria. While discouraged, patients are permitted to continue tobacco use while on the study.
* Age 18 years or older
* ECOG performance status ≤ 2 (Karnofsky ≥60%, see Appendix A)
* Participant must have normal organ and marrow function as defined below within 21 days prior to study registration:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤2.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential (WOCBP) must agree to use appropriate method(s) of contraception. WOCBP should plan to use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 iu/l or equivalent units of hcg) at screening. Pregnancy test will be repeated on the day of the first dose of study drug (before administration), although results of this test are not required for registration.
* "Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception

Exclusion Criteria:

* Known carcinoma in situ (CIS) or invasive squamous cell carcinoma of the oral cavity. A history of a prior stage III (T1-2N1, T3N0) or IV (T1-3N2, T4N0) invasive head & neck squamous cell carcinoma treated with surgery and radiation with or without chemotherapy. Patients with prior locoregionally advanced tumors treated with surgery alone are eligible.
* Existing significant autoimmune conditions. Patients with a history of Hashimoto thyroiditis who are stable on replacement hormone therapy are not excluded. Patients cannot be on long-term (> 4 weeks) corticosteroids at doses exceeding prednisone 20 mg (or its equivalent) prior to enrollment. Short-term corticosteroid dosing is permitted as long as steroids are discontinued within 2 weeks of study registration.
* Subject who has had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Subject who has been treated with immunotherapy. This includes prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known human immunodeficiency virus carrier or a diagnosis of immunodeficiency.
* Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g., Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA is negative).
* A personal history of hematopoietic stem cell or solid organ transplant.
* Known non-infectious pneumonitis or any history of interstitial lung disease.
* A personal history of other active malignancies, with the exception of non-melanomatous skin cancers, low-risk prostate adenocarcinoma on active surveillance, or treated cancers in remission for the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanna GJ, Villa A, Nandi SP, Shi R, ONeill A, Liu M, Quinn CT, Treister NS, Sroussi HY, Vacharotayangul P, Goguen LA, Annino DJ Jr, Rettig EM, Jo VY, Wong KS, Lizotte P, Paweletz CP, Uppaluri R, Haddad RI, Cohen EEW, Alexandrov LB, William WN Jr, Lippman SM, Woo SB. Nivolumab for Patients With High-Risk Oral Leukoplakia: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jan 1;10(1):32-41. doi: 10.1001/jamaoncol.2023.4853. PMID 37971722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Dec 2018 to Jan 2022.
Period: Overall Study
Arm/Group | Nivolumab
Started | 33
Completed | 29
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Progression/Recurrence | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: Years] | 64.7 [32.0 to 79.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  More than one race | 1
  White | 31
ECOG Performance Status (PS) [Count of Participants; unit: Participants] — Measure Description: Eastern Cooperative Oncology Group (ECOG) PS: (PS0) Fully active, able to carry on all pre-disease performance without restriction (PS1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  Participants
    PS 0 | 30
    PS 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR)
Description: BORR on treatment is the percentage of participants who achieved CR or PR. Best overall response is the best response recorded from study registration until the first disease progression/diagnosis of invasive OSCC (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Best overall response was determined by using composite scores based on both measurement and histology, matching to the response grid as following, (1)CR, a decrease of >80% or more; (2)PR, a decrease of 40-80%; (3)SD, neither PR or PD, (4)PD, an increase of 10% or more.
Time Frame: Participants were followed up to 164 days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
percentage of participants | 36.4 [20.4 to 54.9]

2. Secondary Outcome: COMD QLQ Score Change From Baseline to End of Treatment
Description: Quality of Life was evaluated using COMD QLQ (chronic oral mucosal diseases quality of life questionnaire). The range of the possible total score is 0-104, and low score is a good QoL.
Time Frame: Assessed at baseline and end of treatment. Treatment duration in days was a median (range) of 105 (21-164).
Population: This analysis population represents the subset of participants who have completed questionnaires at both baseline and end of treatment.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Nivolumab
Number analyzed (Participants) | 19
Units on a scale | -3 [-36 to 14]
Statistical Analysis 1: Comparison: Nivolumab; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Grade 1/2 Toxicity Rate
Description: The proportion of participants who experienced a maximum grade 1 or 2 adverse events regardless of treatment attribution based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Time Frame: Participants were followed up to 194 days.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
proportion of participants | 0.75 [0.58 to 0.89]

4. Secondary Outcome: Grade 3/4 Toxicity Rate
Description: The proportion of participants who experienced a maximum grade 3 or 4 adverse events regardless of treatment attribution based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Time Frame: Participants were followed up to 194 days.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
proportion of participants | 0.21 [0.09 to 0.39]

5. Secondary Outcome: Time to the Next Surgery for a Head and Neck Malignancy
Description: Time to Next Surgery is defined as time from the first study treatment to any head & neck surgery or resection for biopsy-proven carcinoma in situ (CIS) or invasive oral carcinoma.
Time Frame: Participants were followed up to 13.3 months.
Population: This analysis dataset is comprised of the participants who had next surgery.
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab
Number analyzed (Participants) | 5
Months | 6.5 [2.0 to 13.3]

6. Secondary Outcome: Cancer Free Survival at 2 Years (CFS2)
Description: CFS2 is the probability of participants remaining alive and cancer-free at 2 years based on Kaplan-Meier methodology. Cancer-Free Survival (CFS) is defined as the time from study registration to development of invasive oral cancer or death due to any cause. Participants alive without disease progression or recurrence (of invasive oral cancer) are censored at date of last disease evaluation.
Time Frame: Participants were followed up to 2 years.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
Probability | 0.728 [0.526 to 0.855]

7. Secondary Outcome: 2-year Overall Survival (OS) Rate
Description: 2-year OS rate was defined as the percentage of participants alive at 2 years.
Time Frame: Participants were followed up to 2 years.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
Percentage of participants | 100 [89.4 to 100]

8. Secondary Outcome: PD-L1 Combined Positive Scores (CPS)
Description: PD-L1 CPS (programmed death-1 ligand 1 combined positive score) was calculated by dividing the number of PD-L1 staining cells by the total number of viable tumor cells and then multiplying by 100. Its range of possible values was 0-100, where higher scores were better when participants received PD-L1 targeted therapy.
Time Frame: PD-L1 CPS assessed at baseline.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
score on a scale | 10 [0 to 80]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 2 years; all adverse events were collected up to 194 days
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Per the source vocabulary (CTCAEv4.0) there is a category "Other, specify" for each system organ class. No further data is available to specify classification beyond this general term.
Arm/Group | Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 6/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=33)
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hepatitis viral (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Cardiac troponin T increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=33)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 5
Ear pain (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 7
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 20
Blurred vision (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 2
Floaters (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Periorbital edema (Eye disorders) | 1
Vision decreased (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Oral cavity fistula (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 28
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 3
Immune system disorders - Other, specify (Immune system disorders) | 1
Skin infection (Infections and infestations) | 2
Thrush (Infections and infestations) | 4
Wound infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 12
Cholesterol high (Investigations) | 2
Creatinine increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Thyroid stimulating hormone increased (Investigations) | 1
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Trismus (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2
Genital edema (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 3
Vaginal pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 5
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 14
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT03692325/Prot_SAP_000.pdf